CLINICAL TRIAL: NCT04111159
Title: A Multi-Center, Randomized, Double-Blind, Propofol-Controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of HSK3486 Injectable Emulsion for the Induction of Sedation/Anesthesia in Subjects Undergoing Fiberoptic Bronchoscopy
Brief Title: A Trial Evaluating the Efficacy and Safety of HSK3486 Injectable Emulsion in Subjects Undergoing Fiberoptic Bronchoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK3486-303
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Sedation or Anesthesia
Keywords: Sedation anesthesia fiberoptic bronchoscopy
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): Subjects < 65 years old:0.4mg/kg/0.15mg/kg;Subjects ≥ 65 years old:75% of the dose for subjects < 65 years old.
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): Subjects < 65 years old:2mg/kg/0.75mg/kg;Subjects≥ 65 years old:75% of the dose for subjects < 65 years old.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — Subjects < 65 years old:Initial dose of 0.4 mg/kg followed by 0.15 mg/kg if needed;Subjects ≥ 65 years old:75% of the dose for subjects < 65 years old.
  Arms: HSK3486
Drug: Propofol — Subjects < 65 years old:Initial dose of 2 mg/kg followed by 0.75 mg/kg if needed;Subjects ≥ 65 years old:75% of the dose for subjects < 65 years old.
  Arms: Propofol

SUMMARY:
This is a Multi-Center, Randomized, Double-Blind, Propofol-Controlled Phase III Clinical Trial. Around 260 eligible subjects are planned to be enrolled and randomized in a 1:1 ratio to either the HSK3486 arm or propofol arm. The main objective is to evaluate the efficacy of HSK3486 vs. propofol for the induction of sedation/anesthesia in subjects undergoing fiberoptic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1.Subjects receiving laryngeal mask airway-assisted diagnostic and/or therapeutic fiberoptic bronchoscopy; 2.Male or female, ASA I-III, ≥ 18 and < 80 years old; 3.Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2; 4.Respiratory rate ≥ 10 and ≤ 24 bpm; SpO2 ≥ 93%; SBP ≥ 90 mmHg; DBP ≥ 55 mmHg; HR ≥ 50 and ≤ 100 bpm during screening and baseline periods; 5.Capable of understanding the procedure and method of this study, willing to sign an informed consent form and to complete this study in strict accordance with the study protocol.

-

Exclusion Criteria:

1. Patients with contraindications to deep sedation/general anesthesia or a history of past sedation/anesthesia accidents;
2. Patient known to be allergic to eggs, soy products, opioids and their antidotes, and propofol; patient having contraindications to propofol, opioids and their antidotes;
3. Patients who have undergone endotracheal intubation and/or mechanical ventilation prior to diagnostic or therapeutic bronchoscopy;
4. Medical history or evidence of any of the following prior to screening/at baseline, which may increase sedation/anesthesia risk:

   1. History of cardiovascular diseases: uncontrolled hypertension [systolic blood pressure (SBP) ≥170 mmHg and/or diastolic blood pressure (DBP) ≥105 mmHg without treatment, or SBP > 160 mmHg and/or DBP >100 mmHg after antihypertensive treatment], aneurysm, severe arrhythmia, heart failure, Adams-stokes syndrome, New York Heart Association (NYHA) Class ≥ III, severe superior vena cava syndrome, pericardial effusion, acute myocardial ischemia, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medical treatment, II-III degree atrioventricular block (excluding patients with pacemakers) or QTcF interval ≥ 450 ms [during screening only (corrected using Fredericia's formula1)];
   2. History of respiratory diseases: severe chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, severe airway stenosis, throat mass, history of tracheoesophageal fistula or airway tear, severe respiratory infection within 2 weeks prior to screening;
   3. History of neurological and psychiatric disorders: craniocerebral injury, possible convulsions, intracranial hypertension, cerebral aneurysms, history of cerebrovascular accidents; schizophrenia, mania, insanity, long-term use of psychotropic drugs, and history of cognitive dysfunction;
   4. History of gastrointestinal diseases: gastrointestinal retention, active hemorrhage, or history of gastroesophageal reflux or obstruction that may lead to aspiration;
   5. History of uncontrolled clinically significant liver, kidney, blood system, nervous system or metabolic system diseases judged by the investigator to be probably unsuitable for involvement in the study;
   6. History of alcohol abuse within 3 months prior to screening, abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine);
   7. History of drug abuse within 3 months prior to screening;
   8. History of blood transfusion within 14 days prior to screening;
5. Patients with the following respiratory risks during screening/at baseline:

   1. Acute asthma attack;
   2. Sleep apnea syndrome;
   3. History of malignant hyperthermia or family history;
   4. History of failed tracheal intubation;
   5. Difficult airway (modified Mallampati score ≥ III) as determined by the investigator;
6. Patient who received any of the following medications or treatments during screening/at baseline:

   1. Received any investigational drug within 1 month prior to screening;
   2. Received propofol, other sedatives/anesthetics, and/or opioid analgesics or compounds containing analgesics within 72 h prior to baseline;
7. Laboratory results meeting any of the following criteria during screening/at baseline, confirmed by re-examination:

   1. WBC ≤ 3.0 × 10^9/L;
   2. Platelets ≤ 80 × 10^9/L;
   3. Hemoglobin ≤ 80 g/L;
   4. Prothrombin time ≥ 1.5 × ULN;
   5. Activated partial thromboplastin time (aPTT) ≥ 1.5 × ULN;
   6. ALT and/or AST ≥ 3 × ULN;
   7. Total bilirubin ≥ 1.5 × ULN;
   8. Serum creatinine ≥ 1.5 × ULN.
8. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial; or subjects who are planning pregnancy within 3 month after the completion of the trial (including male subjects);
9. Subject judged by the investigator to have any other factors unsuitable for involvement in the study.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Success rate of fiberoptic bronchoscopy. A successful diagnosis/treatment should meet both of the following: | During induction of sedation/anesthetic on day 1
  1. Completion of fiberoptic bronchoscopy;
  2. No alternative sedation/anesthetic drugs are used, that is, the number of doses of the study drug is ≤ 5 times within any given 15-minute period, starting from the initial administration until the fiberoptic bronchoscopy is completed.

SECONDARY OUTCOMES:
Time to successful sedation/anesthetic induction | From the initial administration of the investigational drug to the first time when MOAA/S is ≤1 on day 1
Time to fully awake | From the last dose of study drug or rescue sedative AND from end of fiberoptic bronchoscopy until the patient has recovered to fully alert on day 1
  the time from the withdrawal of the bronchoscope or the last dose of the study drug to the first of 3 consecutive MOAA/S scores = 5
Time to discharge | Time from the last dose of study drug or rescue sedative and from the end of fiberoptic bronchoscopy until discharge (defined as the ability to walk unassisted) on day 1
  the time from the withdrawal of the bronchoscope or the last dose of the study drug to the first of 3 consecutive Aldrete scores ≥ 9
Use of the investigational drug and alternative drugs | During induction of sedation/anesthetic on day 1
Use of questionnaires to estimate sedation/anesthesia satisfaction, including satisfaction assessments of the subject and anesthesiologist | During induction of sedation/anesthetic on day 1

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, China

REFERENCES:
- [Derived] Luo Z, Tu H, Zhang X, Wang X, Ouyang W, Wei X, Zou X, Zhu Z, Li Y, Shangguan W, Wu H, Wang Y, Guo Q. Efficacy and Safety of HSK3486 for Anesthesia/Sedation in Patients Undergoing Fiberoptic Bronchoscopy: A Multicenter, Double-Blind, Propofol-Controlled, Randomized, Phase 3 Study. CNS Drugs. 2022 Mar;36(3):301-313. doi: 10.1007/s40263-021-00890-1. Epub 2022 Feb 14. PMID 35157236